CLINICAL TRIAL: NCT01010386
Title: A Prospective, Randomized, Double-Blind, Controlled Clinical Trial of the Effects of Oxygen Tension on Clinical In Vitro Fertilization Outcomes
Brief Title: The Effects of Physiologic Oxygen Tension on Clinical In Vitro Fertilization Outcomes
Acronym: PhOx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Pennsylvania (Other); University of California, San Francisco (Other); University of Connecticut (Other)
Responsible Party: Principal Investigator, Heping Zhang, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMN-PhOx
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy; Infertility
Keywords: Pregnancy; Infertility; Physiologic Oxygen Tension; Atmospheric Oxygen Tension
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atmospheric (20%) oxygen tension (Placebo Comparator): Couples will have their gametes and embryos placed in the currently widely used atmospheric (20%) oxygen atmosphere
  Interventions: Procedure: Atmospheric oxygen tension
- physiologic (5%) oxygen tension (Active Comparator): Couples will have their gametes and embryos placed in a physiologic (5%) oxygen atmosphere
  Interventions: Procedure: Physiologic oxygen tension

INTERVENTIONS:
Procedure: Atmospheric oxygen tension — Couples will have their gametes and embryos placed in the currently widely used atmospheric (20%) oxygen atmosphere
  Arms: atmospheric (20%) oxygen tension
Procedure: Physiologic oxygen tension — Couples will have their gametes and embryos placed in a physiologic (5%) oxygen atmosphere
  Arms: physiologic (5%) oxygen tension

SUMMARY:
Primary Aim

* Evaluate whether human embryo exposure to physiologic levels of oxygen during culture improves the percentage of women who deliver a baby following in vitro fertilization and embryo transfer.

Hypothesis to be tested: Physiologic oxygen tension during embryo culture, which approximates the oxygen tension in the fallopian tube and uterus, improves live birth rate in clinical In Vitro Fertilization Embryo Transfer (IVF-ET).

Secondary Aims

Evaluate whether human embryo exposure to physiologic levels of oxygen during culture during in vitro fertilization and embryo transfer

* improves embryo cleavage
* improves clinical pregnancy rate
* reduces multiple pregnancy rate
* reduces miscarriage rate

Hypothesis to be tested: Physiologic oxygen tension during embryo culture, which approximates the oxygen tension in the fallopian tube and uterus, improves embryo cleavage and clinical pregnancy rates and reduces miscarriage rates in clinical IVF-ET.

DETAILED DESCRIPTION:
Study Design

This will be a multi-center, prospective, double-blind clinical trial of physiologic (5%) oxygen tension in culture media vs. standard of care, atmospheric (SOC, 20%) oxygen tension with 840 eligible couples recruited to participate. The randomization scheme will be coordinated through the central data coordinating center (DCC-Yale) and the randomization will be stratified by age group of the woman (18-34, 35-37, 38-40 and 40-42) and each participating site.

Treatment

Couples will be randomized to either have their gametes and embryos placed in a physiologic (5%) oxygen atmosphere or in the currently widely used atmospheric (20%) oxygen atmosphere.

ELIGIBILITY:
Inclusion Criteria:

The critical inclusion criteria will be the diagnosis of infertility and the need for in vitro fertilization as determined by the treating clinician. (We do not plan to alter the standard of care for the indication for IVF at any of the sites.)

* Couple's age must be between 18 and 42 years old
* Patient and partner are scheduled to undergo in vitro fertilization for treatment of infertility
* Couple able to participate in a research project and A) Able to understand study requirements B) Willing to sign informed consent C) Able to return for required follow-up D) Have access to telephone

Exclusion Criteria:

Critical exclusion criteria for this trial will be medical conditions which may complicate treatment or no plans to undergo embryo transfer, as in patients banking embryos prior to cancer therapy. In addition, donor egg and frozen embryo transfer cycles will be excluded.

* Medical contraindication to egg retrieval or pregnancy
* Inability to participate in a research project (Non-English speaking or unable to read or write and/or concurrent participation in any other interventional trial)
* Couple with more than three previous failed IVF cycles
* Donor egg and frozen embryo transfer cycles

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 851 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is live birth rate. | 2 years

SECONDARY OUTCOMES:
The impact of treatment on embryo cleavage | 2 years
The impact of treatment on clinical pregnancy | 2 years
The impact of treatment on multiple pregnancy | 2 years
The impact of treatment on miscarriage | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, MPH, Study Chair — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Director — Albert Einstein College of Medicine; Christos Coutifaris, MD, PhD, Principal Investigator — University of Pennsylvania; Marcelle Cedars, MD, Study Director — University of California, San Francisco; John Nulsen, MD, Study Director — University of Connecticut
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - University of Connecticut, Storrs, Connecticut
  - University of Pennsylvania, Philadelphia, Pennsylvania